CLINICAL TRIAL: NCT06346821
Title: Optimizing Tumor Treating Fields Intervention Timing for Newly Diagnosed Glioblastoma: Insights From Two Emulated Trials With Chinese Multi-Hospital Based Real-World Data
Brief Title: Tumor Treating Fields for Newly Diagnosed Glioblastoma: Two Emulated Trials With Chinese Multi-Hospital Based Real-World Data
Status: Completed | Type: Observational
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhongzheng Xiang, Principal Investigator, Sichuan University
Other Study IDs: WestChinaGBMTTFieldsV1.0
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma; Tumor Treating Fields; Real-world; Concomitant; Adjuvant; Overall survival
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- TTFields-Total: Patients receive standard RT + TMZ, followed by maintenance TMZ, with Optune® starts during peri-radiotherapy period (2 month before to 3 months after radiotherapy). The duration of TTFields lasts for at least 2 months.
  Interventions: Device: Optune® (Tumor Treating Fields)
- Active Comparator: Temozolomide alone: Patients receive RT and TMZ alone, followed by maintenance TMZ.
- TTFields-concomitant: Patients receive TTFields at 200 kHz to the brain using the Optune® System together with RT and TMZ, followed by maintenance TMZ concomitant with the Optune® treatment. The duration of TTFields lasts for at least 2 months. If the subject is assigned to this treatment arm, Optune® therapy will begin no later than the 7th day of RT and TMZ treatment.
  Interventions: Device: Optune® (Tumor Treating Fields)
- TTFields-adjuvant: Patients receive RT and TMZ alone, followed by maintenance TMZ concomitant with TTFields at 200 kHz to the brain using the Optune® within 3 months after radiotherapy for at least 2 months.
  Interventions: Device: Optune® (Tumor Treating Fields)

INTERVENTIONS:
Device: Optune® (Tumor Treating Fields) — TTFields at 200 kHz to the brain using the Optune® System
  Groups: TTFields-Total; TTFields-adjuvant; TTFields-concomitant

SUMMARY:
The goal of this observational study is to learn about the effectiveness of Optune® (Tumor Treating Fields) in newly diagnosed glioblastoma (GBM) in China. The main question it aims to answer are:

* The efficacy of Optune® as an concomitant/adjuvant to radiation therapy (RT) and temozolomide (TMZ) alone in the treatment of newly diagnosed GBM patients.
* The effectiveness of Optune® given concomitantly with RT and TMZ in newly diagnosed GBM patients, compared to RT and TMZ alone.

Participants will:

* Receive or not receive TTFields.
* Concomitantly or adjuvantly receive TTFields.

DETAILED DESCRIPTION:
The goal of this observational study is to learn about the effectiveness of Optune® (Tumor Treating Fields) in newly diagnosed glioblastoma (GBM) in China. The main question it aims to answer are:

* The efficacy of Optune® as an concomitant/adjuvant to radiation therapy (RT) and temozolomide (TMZ) alone in the treatment of newly diagnosed GBM patients.
* The effectiveness of Optune® given concomitantly with RT and TMZ in newly diagnosed GBM patients, compared to RT and TMZ alone.

Participants will:

Step 1:

* Treatment arm I: Patients receive standard RT + TMZ, followed by maintenance TMZ, with Optune® starts during peri-radiotherapy period (2 month before to 3 months after radiotherapy). The duration of TTFields lasts for at least 2 months.
* Treatment arm II: Patients receive RT and TMZ alone, followed by maintenance TMZ concomitant.

Step 2:

* Treatment arm I: Patients receive TTFields at 200 kHz to the brain using the Optune® System together with RT and TMZ, followed by maintenance TMZ concomitant with the Optune® treatment. The duration of TTFields lasts for at least 2 months. If the subject is assigned to this treatment arm, Optune® therapy will begin no later than the 7th day of RT and TMZ treatment.
* Treatment arm II: Patients receive RT and TMZ alone, followed by maintenance TMZ concomitant with TTFields at 200 kHz to the brain using the Optune® within 3 months after radiotherapy for at least 2 months.

Researchers will compare the overall survival of each arm to see if TTFields demonstrates an improvement in survival outcomes within the Chinese population in real-world practice, and whether this efficacy is further enhanced when combined with RT and TMZ.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of GBM according to WHO classification criteria.
2. Age ≥ 18 years.
3. Recovered from maximal debulking surgery.
4. Karnofsky performance status ≥ 60.
5. Planned treatment with RT/TMZ followed by maintenance TMZ.

Exclusion Criteria:

1. Progressive disease (per investigator's assessment).
2. Infratentorial or leptomeningeal disease.
3. Significant co-morbidities at baseline which would preclude maintenance RT or TMZ treatment.
4. Any serious surgical/post-operative condition that may risk the patient according to the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are diagosed and whose surgery and radiotheraoy are finished in West China Hospital, Sichuan Cancer Hospital, Shenzhen People's Hospital, Henan Cancer Hospital, The First Affiliated Hospital of Xi'an Jiaotong University, The First Affiliated Hospital of Zhengzhou University
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | 5 years
  Survival will be measured from the time of randomization until date patient is alive.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Liu, PhD, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, Analytic Code